CLINICAL TRIAL: NCT06759324
Title: Randomized Controlled Pilot Clinical Study Including Kombucha in the Diet of Individuals with Overweight and Class 1 Obesity: Comparative Assessment Between Live and Pasteurized Kombucha and Its Effects on Gut Microbiota, Metabolic Parameters, and Liver Function [FUSILLI Project -H2020]
Brief Title: Kombucha in Overweight and Obese: Live Vs. Pasteurized Effects on Microbiota, Metabolism, and Liver Function
Acronym: KOMBIOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associação Centro de Apoio Tecnológico Agro Alimentar (Other)
Responsible Party: Principal Investigator, Inês Brandão, Principal Investigator, Associação Centro de Apoio Tecnológico Agro Alimentar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FUSILLI: PARECER (02/2024); Grant agreement No. 101000717 (Other Grant/Funding Number: European Union's Horizon 2020 research and innovation programme)
Record Dates: First submitted 2024-12-09; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity and Overweight
Keywords: kombucha; gut microbiota; obesity; liver function; fermented beverages; Randomized Controlled Trial; overweight; fermented tea; SCOBY; live vs pasteurized kombucha; Small Intestinal Bacterial Overgrowth (SIBO); Bristol Stool Form Scale; Likert Scale Analysis; Nutritional Interventions; Inflammatory Biomarkers; metabolic parameters
MeSH Terms: conditions — Obesity; Overweight | interventions — Carbonated Water

STUDY DESIGN:
Intervention Model Description: The study aims to recruit at least 30 individuals with overweight and class 1 obesity, aged between 18 and 60 years, randomly distributed into 3 arms (each arm should have about 10 participants). The first arm receives a daily amount of 33 cl of kombucha (live drink) for 4 weeks, the second arm receives a daily amount of 33 cl of kombucha (pasteurized drink) for 4 weeks. The control group receives 33 cl of water for 4 weeks. Kombucha samples are prepared for the study by Erfrischerling GmbH & Co. KG (Germany).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Partial double blinding (participants will not know if they are consuming live or pasteurized kombucha; the nutritionist will not know which arm the participant belongs to; the technician responsible for microbiota sequencing will receive coded samples without information regarding the intervention/control arm the sample belongs to).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention: Kombucha (live drink) (Experimental): The first arm receives a daily amount of 33 cl of kombucha (live drink) for 4 weeks (dietary supplement).
  Interventions: Dietary Supplement: Live kombucha (non filtered/ non pasteurized)
- Intervention: Pasteurized kombucha (Experimental): The second arm receives a daily amount of 33 cl of kombucha (pasteurized drink) for 4 weeks (dietary supplement).
  Interventions: Dietary Supplement: Pasteurized kombucha (non filtered)
- Sparkling water (Active Comparator): The third arm receives 33 cl of sparkling water for 4 weeks (control).
  Interventions: Other: Control (sparkling water)

INTERVENTIONS:
Dietary Supplement: Live kombucha (non filtered/ non pasteurized) — Participants receive a daily amount of 33 cl of live kombucha (non-pasteurized/ non-filtered) for 4 weeks (28 days).
  Arms: Intervention: Kombucha (live drink)
Dietary Supplement: Pasteurized kombucha (non filtered) — Participants receive a daily amount of 33 cl of kombucha (pasteurized drink) for 4 weeks (28 days).
  Arms: Intervention: Pasteurized kombucha
Other: Control (sparkling water) — Participants receive a daily amount of 33 cl of sparkling water for 4 weeks.
  Arms: Sparkling water

SUMMARY:
Kombucha, a fermented beverage made from Camellia sinensis tea (black, oolong, or green) with sugar and a symbiotic culture of bacteria and yeast (SCOBY), has gained global attention for its potential health benefits. Factors like the type and amount of sugar substrate, fermentation time, and temperature significantly influence its organic compounds, total phenolics, vitamin content, and alcohol levels.

In a previous study, kombucha's impact on glucose tolerance, insulin sensitivity, body composition, and liver function was tested in male prediabetic mice with diet-induced obesity. Daily supplementation (200 µL per mouse) improved glucose tolerance after nine days (equivalent to one year in humans) and reduced liver steatosis, despite no changes in body composition.

Although kombucha has been associated with antioxidant, antimicrobial, probiotic, antidiabetic, and anticancer activities, strong scientific evidence in humans remains limited. Further clinical studies are needed to substantiate kombucha's health benefits in humans.

DETAILED DESCRIPTION:
The objectives of this clinical study aim to explore the effects of kombucha on the health of individuals with overweight and class 1 obesity, while also determining whether the kombucha microbiota plays a role in the observed effects. Specifically, by investigating metabolic parameters such as glucose and insulin levels and lipid profile, as well as the composition and diversity of the gut microbiota and liver function, the study will contribute to a deeper understanding of the potential benefits and mechanisms of action of kombucha consumption in humans. The study aims to recruit at least 30 individuals with overweight and class 1 obesity, aged between 18 and 60 years, randomly distributed into 3 arms (each arm should have about 10 participants). The first arm receives a daily amount of 33 cl of kombucha (live drink) for 4 weeks, the second arm receives a daily amount of 33 cl of kombucha (pasteurized drink) for 4 weeks. The control group receives 33 cl of sparkling water for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

Individuals with a Body Mass Index (BMI) between 25 kg/m² and 34.9 kg/m², of both biological sexes, aged between 18 and 60 years, available to comply with the study protocol (described in this document) and sign informed consent.

Exclusion Criteria:

Volunteers will be excluded from the study if they present one or more of the following conditions:

1. Subjects with sensitivity to kombucha;
2. Consumption of kombucha, kefir, kimchi, cheese, raw vinegar, sauerkraut, kvass, and other fermented products during the study and in the 3 weeks before the study.
3. Use of antibiotics in the 6 months prior to the start of the study;
4. Use of pro/prebiotics or fibers as dietary supplements or any food/molecule that modifies intestinal transit time 6 weeks before recruitment; use of laxatives 6 weeks before recruitment;
5. Specific dietary regimen (e.g., vegan); specific dietary treatment (e.g., high protein);
6. Excessive consumption of substances and alcohol; smokers;
7. Diagnosis of gastrointestinal disorders, hormonal or thyroid diseases, autoimmune diseases, and/or chronic use of corticosteroids; psychiatric disease; Type 1 or 2 diabetes;
8. Use of proton pump inhibitors; antidiabetic drugs or insulin and statins;
9. Subjects with insulin sensitivity;
10. Pregnant or lactating women;
11. Subjects with tooth sensitivity
12. Participation in another clinical trial in the last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Gut microbiota composition and diversity (fecal samples) | 4 weeks
  Analyze the changes in the relative abundance of the microbial species present, including taxonomic identification and diversity analysis, from baseline to the end of intervention, by next-generation sequencing (NGS).
Change in fasting glucose levels | 4 weeks
  Fasting glucose (mg/dl), from baseline to the end of intervention. Reduction is a better outcome.
Change in fasting insulin levels | 4 weeks
  Fasting insulin (μUI/mL), from baseline to the end of intervention. Reduction is a better outcome.
Changes in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) values | 4 weeks
  HOMA-IR values, from baseline to the end of intervention. Calculated from fasting glucose (mmol/L) X fasting insulin (mU/L) / 22.5). Less than 1.0 means insulin-sensitive, which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance. Reduction is a better outcome.
Changes in Lipid profile | 4 weeks
  Lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides), in mg/dL, from baseline to the end of intervention.

SECONDARY OUTCOMES:
Stool consistency rating by Bristol Stool Scale | 4 weeks
  The Bristol Stool Chart is a medical tool used to classify human feces into seven distinct categories. This scale is widely regarded as the gold standard for evaluating stool consistency and intestinal transit time in adults. It ranges from type 1 (separate hard lumps), which indicates the slowest transit time and constipation, to type 7 (watery with no solid pieces), representing the fastest transit time. Daily monitoring questionnaire (to evaluate 1 to 7), from baseline to the end of intervention.
Variation in SIBO diagnosis (positive/negative) measured by methane and hydrogen levels in breath test | 4 weeks
  Hyrogen and methane lactulose breath test, in ppm, from baseline to end of intervention. Interpretation criteria: SIBO test is positive if there is an early increase (in the first 90 minutes) equal to or greater than 20 ppm of H2 and/or equal to or greater than 10 ppm of CH4, when compared with the lowest value obtained.
Change in liver enzyme levels | 4 weeks
  Analyze liver enzymes (units: in UI/L) such as alkaline phosphatase, alanine transaminase, aspartate transaminase, gamma-glutamyl transferase, from baseline to end of intervention, to determine potential hepatic effects of Kombucha consumption.
Change in levels of oxidative stress biomarker (ratio 8-iso-PGF2α to prostaglandin F2α (PGF2α)) | 4 weeks
  Measure of oxidative stress biomarker (pg/mL ), from baseline to the end of intervention. Normal human plasma reference values: 40-100 pg/mL.
Change in gastrointestinal symptoms using a Likert scale | 4 weeks
  Evaluate gastrointestinal symptoms (e.g., bloating, gas) using a 10-point Likert scale, from baseline to the end of intervention. The daily questionnaire goes from zero (0) which means "no pain" to ten (10) which means "worst pain imaginable".
Change in high-sensitive C-reactive protein levels | 4 weeks
  Levels of h-sensitivity C-reactive protein (hsCRP), a marker of inflammation, in mg/dL, from baseline to the end of intervention. hsCRP levels of less than 0.100, 0.100 to 0.300, and greater than 0.301 mg/dL are associated with lower, moderate, and higher cardiovascular risks, respectively.
Change in Total oxidant capacity | 4 weeks
  Oxidative stress biomarker, pg/mL, measured from baseline to the end of intervention. Normal values range from 40-100.
Changes in serum albumin and bilirubin levels | 4 weeks
  Evaluate hepatobiliary function, albumin (g/dL), Bilirubin (mg/dL)
Changes in short chain fatty acids in stool | 4 weeks
  SCFAs in stool, units µM

OTHER OUTCOMES:
Body weight change | 4 weeks
  Anthropometric measurement, unit of measure: Kg
BMI change | 4 weeks
  Body mass index (BMI) is a measure of body fat based on height and weight, unit of measure: Kg/m2
Waist circumference change | 4 weeks
  Anthropometric measurement, unit of measure: cm
Body fat percentage change | 4 weeks
  unit of measure: %
Changes in kidney function biomarkers- creatinin, urea and uric acid | 4 weeks
  units in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Brandão, PhD, Principal Investigator — CATAA
Locations (2):
- Portugal (2):
  - Centro de Apoio Tecnológico Agro Alimentar (CATAA), Castelo Branco, Castelo Branco District
  - Centro de Apoio Tecnológico Agro Alimentar (CATAA) (facilities temporarily provided by the Affidea clinical analysis center), Covilha

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreira GV, Araujo LCC, Murata GM, Matos SL, Carvalho CRO. Kombucha tea improves glucose tolerance and reduces hepatic steatosis in obese mice. Biomed Pharmacother. 2022 Nov;155:113660. doi: 10.1016/j.biopha.2022.113660. Epub 2022 Sep 12. PMID 36095960